CLINICAL TRIAL: NCT05923814
Title: The Administration of Humanized Anti-CD25 Antibody for Prophylaxis of aGVHD in Patients Older Than 50y Underwent HID-HSCT
Brief Title: Humanized Anti-CD25 Antibody for Prophylaxis of aGVHD in Elderly Underwent HID-HSCT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-CD25-01-CAMS
Record Dates: First submitted 2023-06-20; First posted 2023-06-28 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-05

CONDITIONS: The Effecacy and Safety of Humanized CD25 Antibody in aGVHD Prophylaxis Among Elderly Patients After HID-HSCT

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- treatment arm (Experimental)
  Interventions: Drug: CD25 prophylaxis

INTERVENTIONS:
Drug: CD25 prophylaxis — The humanized CD25 antibody was administered at 1 mg/kg iv on days+1 and +4 after HSCT.

SUMMARY:
Age is no longer a barrier to successful allogeneic hematopoietic cell transplantation. However, the incidence of aGVHD is still high among the elderly, especially for patients receiving HID-HSCT. We designed this clinical trial to use humanized CD25 antibody for aGVHD prophylaxis among in elderly patients aged 50 and older. The humanized CD25 antibody was administered at 1 mg/kg iv on days+1 and +4 after HSCT.

ELIGIBILITY:
Inclusion Criteria:

* (1) hematological malignances patients underwent HLA-haploidentical donor HSCT. (2) Age elder than or equal to 50 years; (3) Informed consent may be signed by themselves. (4) HIV negative, HBV, HCV negative; (5) Informed consent must be signed before the start of the study procedures, and informed consent must be signed by the patient himself or his immediate family. Considering the patient 's condition, if the patient' s signature is unfavorable for disease treatment, the informed consent form should be signed by the legal guardian or the patient 's immediate family member.

Exclusion Criteria:

* (1) received a previous allogeneic HSCT; (2) Uncontrolled infection at enrollment; requires mechanical ventilation or is hemodynamically unstable at the time of enrollment; (3) has severe hepatic insufficiency (defined as Child-Pugh Class C; has serum aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 5 xthe upper limit of normal (ULN) or serum total bilirubin > 2.5 x ULN.

  (4) has end-stage renal impairment with a creatinine clearance less than 10 mL/min.

  (5) has both moderate hepatic insufficiency AND moderate renal insufficiency; (6) has documented positive results for human immunodeficiency virus antibody (HIVAb), hepatitis C virus antibody (HCV-Ab) with detectable HCV RNA, or hepatitis B surface antigen (HBsAg) within 90 days prior to enrollments; (7) has active solid tumor malignancies with the exception of localized basal cell or squamous cell skin cancer or the condition under treatment (e.g., lymphomas).

  (8) Suffering from mental disorders or other conditions and unable to cooperate with the requirements of study treatment and monitoring; (9) unable or unwilling to sign the consent form; (10) patients with other special conditions assessed as unqualified by the investigator

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-07-07 (Estimated); Primary Completion 2024-05-07 (Estimated); Study Completion 2024-05-07 (Estimated)

PRIMARY OUTCOMES:
the incidence of aGVHD | 24 weeks after HSCT